CLINICAL TRIAL: NCT06041425
Title: The Effects of Single Dose Oxycodone Versus Sufentanil on Pain and Inflammatory Response After Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma: a Randomized Controlled Study
Brief Title: The Effects of Oxycodone Versus Sufentanil on Pain and Inflammatory Response After TACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-SR-093
Record Dates: First submitted 2023-08-09; First posted 2023-09-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma; Transcatheter Arterial Chemoembolization; Pain; Inflammation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pain; Inflammation | interventions — Oxycodone; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxycodone (Experimental): The patients were given 0.1mg/kg oxycodone 15 minutes before transcatheter arterial chemoembolization (TACE).
  Interventions: Drug: Oxycodone
- Sufentanil (Active Comparator): The patients were given 0.1μg/kg sufentanil 15 minutes before transcatheter arterial chemoembolization (TACE).
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Oxycodone — The patients were given 0.1mg/kg oxycodone 15 minutes before transcatheter arterial chemoembolization (TACE). WBC count, neutrophil percentage, CRP, and IL-6 were used as inflammatory markers and measured before TACE (1 day before TACE) and 24 hours after TACE. Assess pain and side effects during TACE and within 24 hours after TACE. Pain was evaluated using the 11 point Numeric Rating Scale (NRS).
  Other Names: preemptive analgesia
  Arms: Oxycodone
Drug: Sufentanil — The patients were given 0.1μg/kg sufentanil 15 minutes before transcatheter arterial chemoembolization (TACE). WBC count, neutrophil percentage, CRP, and IL-6 were used as inflammatory markers and measured before TACE (1 day before TACE) and 24 hours after TACE. Assess pain and side effects during TACE and within 24 hours after TACE. Pain was evaluated using the 11 point Numeric Rating Scale (NRS).
  Other Names: preemptive analgesia
  Arms: Sufentanil

SUMMARY:
The purpose of this randomized, double-blind trial was to compare the effects of preemptive Oxycodone and sufentanil at the same dose on pain and inflammatory response after transcatheter arterial chemoembolization (TACE) of hepatocellular carcinoma. To study the effect of single dose intravenous injection of Oxycodone and sufentanil before TACE on inflammatory reaction after TACE; And (ii) evaluate the effects of different opioid drugs on pain and nausea/vomiting after TACE.

DETAILED DESCRIPTION:
Transcatheter arterial chemoembolization (TACE) is currently considered as the treatment for unresectable hepatocellular carcinoma (HCC). Due to sudden blockage of the main blood vessels supplying the tumor, local liver tissue swells and the tumor rapidly necroses. A large number of inflammatory mediators, including white blood cell (WBC) count, C-reactive protein (CRP) and Interleukin 6 (IL-6), will inevitably appear in TACE induced ischemic and/or necrotic tissue reactions, which contribute to the development of pain. Pain can worsen the patient's quality of life, prolong hospital stay, and increase costs. 93% of patients require opioid therapy during and after TACE.

Opioids are the most common drugs for treating pain. There are three types of opioid receptors, μ Receptors κ Receptors and δ Receptors. Sufentanil is a highly selective drug μ Receptor agonists have fast onset and strong analgesic effects. However, sufentanil is not as effective as Oxycodone in relieving visceral pain. Oxycodone not only activates μ receptors, also occupying κ receptors, alleviate visceral ischemic pain and inflammatory reactions.

In addition to the type of medication, the administration time can also affect perioperative pain. Preemptive analgesia refers to the intervention of pain relief before nociceptive stimuli to suppress the progression of stress states and central sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Presence of histologically confirmed or clinically diagnosed hepatocellular carcinoma (fulfilling the criteria for lesions with typical imaging);
* Presence of Child-Pugh class A or B disease;
* Absence of benefit from a treatment of established efficacy such as resection and local ablation;
* ECOG:0-2.

Exclusion Criteria:

* Extrahepatic metastasis and/or microvascular invasion;
* Severe liver and kidney dysfunction;
* Uncontrolled or significant cardiovascular disease; Autoimmune hepatitis; Long term use of opioids, steroid hormones, and non steroidal anti-inflammatory drugs; Abnormal elevation of C-reactive protein (CRP); Increased white blood cells (>11000/mm3); Study Drugs allergy; Patients who were treated within 4 weeks after COVID-19 infection was diagnosed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Intraoperative pain intensity during TACE. | Intraoperative (From the beginning of TACE to the end of TACE.)
  Pain intensity is assessed by numerical rating scale pain scores (0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome).
Pain intensity at 1hour after the end of TACE. | From 0 to 1 hour after the end of TACE.
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome).
Pain intensity at 6hours after the end of TACE. | From 1hour to 6 hours after the end of TACE.
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome).
Pain intensity at 12hours after the end of TACE. | From 6hours to 12 hours after the end of TACE.
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome).
Pain intensity at 24hours after the end of TACE. | From 12 hours to 24 hours after the end of TACE.
  Pain intensity is assessed by numerical rating scale pain scores(0-10,0 represents painless,10 represents intolerable pain;higher scores mean a worse outcome).

SECONDARY OUTCOMES:
The WBC count | 24 hours
  The WBC count in 10^9/L. Inflammatory reactions
Neutrophil percentage | 24 hours
  neutrophil percentage in %.
  Inflammatory reactions
Level of CRP | 24 hours
  CRP in mg/L.
  Inflammatory reaction
Level of IL-6 | 24 hours
  IL-6 in pg/mL.
  Inflammatory reaction
Nausea and vomiting scale | 24 hours
  Nausea and vomiting were graded on a four-point scale, 0,no nausea.1,mild nausea. 2,severe nausea requiring antiemetics. and 3, retching and/or vomiting.)

CONTACTS AND LOCATIONS:
Overall Officials: Yu CHEN, MD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: August 2023 to August 2024
Access Criteria: Within one year